CLINICAL TRIAL: NCT05809635
Title: Natural History Study in Retinitis Pigmentosa Caused by Mutations in the BEST1 Gene
Brief Title: Study of BEST1 Vitelliform Macular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Universität Tübingen (Other); Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Stephen H. Tsang, Laszlo Z. Bito Professor of Ophthalmology and Professor of Pathology and Cell Biology, Columbia University
Other Study IDs: AAAT5994; R24EY028758 (NIH)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Best Vitelliform Macular Dystrophy; Retinitis Pigmentosa
MeSH Terms: conditions — Vitelliform Macular Dystrophy; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Best Vitelliform Macular Dystrophy (VMD) Participants: Participants with a clinical picture of Retinitis pigmentosa with dominant and recessive variants in the BEST1 gene
  Interventions: Other: Natural History Study

INTERVENTIONS:
Other: Natural History Study — Longitudinal assessment of participants with BEST1 Vitelliform Macular Dystrophy

SUMMARY:
The purpose of this study is to establish the natural history of of participants with BESTROPHIN 1 Vitelliform Macular Dystrophy.

The blinding disorder Best Vitelliform Macular Dystrophy (VMD) is caused by any one of more than 250 different mutations in the BEST1 gene.

As new treatments are developed, a clear understanding of the natural history of disease progression of BEST1 VMD is necessary. The goals of this natural history study are to:

1. Report the natural history of retinal degeneration in participants with a clinical diagnosis of VMD with molecular confirmation of a pathogenic BEST1 mutation(s).
2. Identify sensitive structural and functional outcome measures to use for future multicenter clinical trials for the treatment of BESTROPHIN 1 VMD.
3. Compare progression of the identified structural and functional measures between the two eyes to judge the suitability of the second untreated eye as a control for a future clinical trial involving unilateral treatment
4. Identify well-defined patient populations for future clinical trials of investigative treatments for BEST1 VMD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Diagnosis of BEST1-associated VMD by study physician, who are trained retinal specialists in the university clinic Must be able to commit to 4 follow-up study visits (3 years)

Exclusion Criteria:

* Systemic condition that prevents the participant from undergoing the exams

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are expected to present to the clinic at all age groups; enrollment of subjects <18 years of age will be obtained by informed consent in the company of a parent or legal guardian. There will also be no gender-or ethnic/racial specific inclusion criteria. The enrollment of non-English speaking subjects is not expected.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Medmont Dark Adapted Chromatic (DAC) Automated Perimeter | Up to 3 years
Full-field electroretinogram (ERG) | Up to 3 years
  ERG conducted under International Society for Clinical Electrophysiology of Vision (ISCEV) Protocol.
Electroocoulogram (EOG) | Up to 3 years
  EOG conducted under International Society for Clinical Electrophysiology of Vision (ISCEV) Protocol
Optical Coherence Tomography (OCT) | Up to 3 years
Fundus Autofluorescence (FAF) | Up to 3 years
Near-infrared fundus autofluorescence (NIR-AF) | Up to 3 years
Quantitative Fundus Autofluorescence (qAF) | Up to 3 years

SECONDARY OUTCOMES:
Best-corrected Visual Acuity (BCVA) | Up to 3 years
Color Fundus Photos | Up to 3 years
Macular Integrity Assessment (MAIA) Microperimetry | Up to 3 years
Goldman Kinetic Visual Field | Up to 3 years
Light-adapted Static Perimetry | Up to 3 years
Dark-adapted Chromatic Perimetry | Up to 3 years
Full-field Stimulus Testing | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Tsang, MD, PhD, Principal Investigator — Columbia University
Locations (3):
- Columbia University Irving Medical Center, New York, New York, United States
- Institut de la Vision/Centre de maladies rares du Centre Hospitalier National Ophtalmologique des Quinze-Vingts, Paris, France
- Eberhard Karls University Tubingen, Tübingen, Germany